CLINICAL TRIAL: NCT04595799
Title: MS Screen Test: Using a Smartphone Application to Predict the Prognosis in Patients With Newly Diagnosed Multiple Sclerosis
Brief Title: Use of a Smartphone Application to Predict the Prognosis in Patients With Newly Diagnosed Multiple Sclerosis.
Acronym: MSST
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20-AOI-01
Record Dates: First submitted 2020-10-07; First posted 2020-10-22 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multiple sclerosis (MS) is a chronic demyelinating disease of the central nervous system for which the investigators now have many treatment alternatives. These treatments have a preventive goal and the data in the literature suggest the interest in rapidly achieving optimal control of the disease in order to decrease the risk of long-term disability progression.

One of the current unmet needs is to have markers that can be used at the individual level to predict the long-term prognosis in order to propose optimal and personalized therapeutic management.

Classically used clinical markers do not meet this need. It is recognized that there is a so-called silent course of MS (not measurable by clinical parameters), which may, after several months or years, be expressed as a physical or cognitive disability.

MRI is the reference examination for monitoring the sub-clinical activity of the disease but it does not allow the neurodegenerative side of the disease to be assessed. Other blood or imaging markers are being studied but are not yet usable in daily practice.

The project aims to evaluate the interest in using digital biomarkers, based on a rapid assessment of patients using a locally developed mobile application (MS Screen Test - MSST) to predict the evolutionary prognosis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 60 years of age
* Presenting a diagnosis of relapsing-remitting MS defined according to McDonald 2017 criteria confirmed within 6 months prior to inclusion
* Starting first-line treatment (interferon beta, glatiramer acetate, teriflunomide, dimethyl fumarate)
* Having an encephalic and cervical MRI in OFSEP format, within 6 months prior to inclusion
* No relapse within 30 days prior to inclusion

Exclusion Criteria:

* presence of a motor, visual or cognitive deficit not related to MS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with newly diagnosed multiple sclerosis starting first-line background therapy
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2025-11-09 (Estimated); Study Completion 2025-11-09 (Estimated)

PRIMARY OUTCOMES:
speed test in MMST results | 12 months
  the average speed (in taps per second or Hz) for the dominant and non-dominant hand
agility test in MMST results | 12 months
  time required (in seconds) to bring the ball to the target as well as the actual time the ball will be held inside the target (expressed as a percentage of the total recording time)
synchronization test in MMST results | 12 months
  the average time interval expressed in milliseconds separating the left and right index strokes.
visual test in MMST results | 12 months
  number of letters seen
Cognitive test in MMST results | 12 months
  the average response latency (the time in milliseconds between the display and the click on a good answer) expressed in milliseconds, the number of wrong answers as well as the number of missed letters.
  the average response latency is the combination of multiple measurements (time of response, number of wrong answers and number of missed letters.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Lille University Hospital, Lille
  - LYON Civil Hospital, Lyon
  - Montpellier university hospital, Montpellier
  - Nice University Hospital, Nice
  - Nimes University Hospital, Nîmes
  - Paris University Hospital - la pitié salpétriere, Paris
  - Rennes University Hospital, Rennes
  - Rouen University hospital, Rouen
  - Strasbourg University Hospital, Strasbourg
  - Toulouse university hospital, Toulouse